CLINICAL TRIAL: NCT03489837
Title: A Randomized, Double-blind, Multicenter, Active-controlled Phase III Study to Evaluate the Efficacy and Safety of Levotuss CR Tab. in Comparison With Levotuss Syrup in Patients With Cough Due to Acute or Chronic Bronchitis
Brief Title: Phase III Study to Evaluate the Efficacy and Safety of HOB-048 CR Tab. in Comparison With HOB-048 Syrup in Patients With Cough Due to Acute or Chronic Bronchitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hyundai Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOB-048
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Evaluate the Efficacy and Safety of Levotuss CR Tab. in Comparison With Levotuss Syrup in Patients With Cough Due to Acute or Chronic Bronchitis
MeSH Terms: conditions — Bronchitis, Chronic | interventions — dipropizine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levotuss CR tab (Experimental): oral taken
  Interventions: Drug: Levotuss
- Levotuss syrup (Active Comparator): oral taken
  Interventions: Drug: Levotuss

INTERVENTIONS:
Drug: Levotuss — oral taken

SUMMARY:
A randomized, double-blind, multicenter, active-controlled phase III study to evaluate the efficacy and safety of Levotuss CR tab. in comparison with Levotuss syrup in patients with cough due to acute or chronic bronchitis

ELIGIBILITY:
Inclusion Criteria:

* moderate, severe, very severe non-productive cough patients

Exclusion Criteria:

* Patients receiving a concomitant therapy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Cough severity check | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Included Seoul national hospital,10sites, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes